CLINICAL TRIAL: NCT01553331
Title: Day Case Laparoscopic Cholecystectomy: Comparison of Fundus First With Ultrasonic Dissection or Conventional Diathermy Hook, Randomized Trial
Brief Title: Day Case Laparoscopic Cholecystectomy: Fundus First With Ultrasonic Dissection or Conventional Diathermy Hook
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Anne Mattila, MD, Central Finland Hospital District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSSHPB10208
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Cholecystolithiasis
Keywords: laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystolithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional diathermy hook (Active Comparator): Laparoscopic cholecystectomy made with diathermy hook starting from Calot´s triangle
  Interventions: Procedure: dissection of gallbladder in laparoscopic cholecystectomy
- ultrasonic dissection (Active Comparator): Laparoscopic cholecystectomy made with ultrasonic dissection starting from gallbladder fundus
  Interventions: Procedure: dissection of gallbladder in laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: dissection of gallbladder in laparoscopic cholecystectomy — Laparoscopic cholecystectomy with diathermy hook starting from triangle of Calot
  Arms: conventional diathermy hook
Procedure: dissection of gallbladder in laparoscopic cholecystectomy — laparoscopic cholecystectomy with ultrasonic scissors starting from fundus
  Arms: ultrasonic dissection

SUMMARY:
Day case laparoscopic cholecystectomy can be made with conventional diathermy hook starting at triangle of Calot´s. Ultrasonic dissection starting from the gallbladder fundus is another option. The aim is to test the hypothesis that with ultrasonic dissection technique a better same day discharge and a shorter operative time can be achieved.

DETAILED DESCRIPTION:
After initiation of general anesthesia patients are randomized either to conventional or ultrasonic dissection group. The patients and recovery room personnel are blinded to the operative technique used.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* BMI under 35
* normal liver enzymes
* no bile duct dilatation in ultrasound
* cholecystolithiasis

Exclusion Criteria:

* NSAID allergy
* previous upper gi-surgery
* common bile duct stones in preoperative imaging
* history of severe acute pancreatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
same day discharge | 30 days
operative time | 30 days
intraoperative complications | 30 days

SECONDARY OUTCOMES:
analgetic use | 30 days
postoperative nausea and vomiting | 30 days
readmission | 30 days
morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ilmo Kellokumpu, Docent, Study Director — Jyvaskyla Central Hospital; Anne K Mattila, MD, Principal Investigator — Jyvaskyla Central Hospital
Locations (1):
- Jyvaskyla Central Hospital, Jyväskylä, Jyvaskyla, Finland

REFERENCES:
- [Background] Cengiz Y, Janes A, Grehn A, Israelsson LA. Randomized trial of traditional dissection with electrocautery versus ultrasonic fundus-first dissection in patients undergoing laparoscopic cholecystectomy. Br J Surg. 2005 Jul;92(7):810-3. doi: 10.1002/bjs.4982. PMID 15880649
- [Background] Cengiz Y, Dalenback J, Edlund G, Israelsson LA, Janes A, Moller M, Thorell A. Improved outcome after laparoscopic cholecystectomy with ultrasonic dissection: a randomized multicenter trial. Surg Endosc. 2010 Mar;24(3):624-30. doi: 10.1007/s00464-009-0649-2. Epub 2009 Aug 18. PMID 19688393